CLINICAL TRIAL: NCT03398694
Title: A Phase II Study Analyzing Pre-operative Stereotactic Radiosurgery Followed by Resection for Patients With 1 - 4 Brain Metastases
Brief Title: Pre-operative Stereotactic Radiosurgery Followed by Resection for Patients With Brain Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Namita Agrawal, Assistant Professor of Radiation Oncology, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0627; 1707314702 (Other: Indiana University IRB)
Record Dates: First submitted 2018-01-08; First posted 2018-01-12 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): This is a single arm study so this arm will include all eligible subjects. All subjects will have radiosurgery 1-4 days prior to surgical resection.
  Interventions: Procedure: Radiosurgery

INTERVENTIONS:
Procedure: Radiosurgery — Stereotactic radiosurgery will be delivered on all patients utilizing gamma knife or linear accelerator based techniques as per RTOG-9005 dosing criteria (Section 11 Table 1) based on tumor diameter with the exception that the largest lesion diameter to be treated with 15 Gy will be 5 cm. All apparent, previously untreated brain metastases will be treated with radiosurgery at this time.
  Radiosurgery will be performed 1-4 days prior to surgical resection. Vital signs and MRI Brain planning scan will be performed on the day of radiosurgery prior to the procedure.

SUMMARY:
This is a prospective, single arm, phase II trial to determine the local control at 6 months utilizing pre-operative stereotactic radiosurgery followed by surgery within 1 - 4 days in subjects with a diagnosis of 1-4 brain metastases and with an indication for surgical resection of at least one brain metastasis at the discretion of a neurosurgeon.

DETAILED DESCRIPTION:
Primary Objective To evaluate 6 month in-brain local control utilizing pre-operative stereotactic radiosurgery followed by surgical resection for brain metastases.

Secondary Objectives

* Overall survival
* Distant in-brain progression
* Rate of leptomeningeal spread
* Rate of radiation necrosis

ELIGIBILITY:
Inclusion Criteria

1. Radiographically confirmed solid tumor brain metastases
2. Criteria for surgical resection of at least one metastasis per neurosurgeon discretion
3. A diagnostic MRI Brain or CT Head demonstrating the presence of 1-4 solid tumor brain metastases and lesion to be resected no more than 5 cm in any direction, performed within 30 days prior to stereotactic radiosurgery. If multiple lesions are present, then the total brain metastases volume can be no more than 30 cm3 excluding the lesion to be resected.
4. For known primary included in brainmetgpa.com, an estimated median survival no less than 6 months per brainmetgpa.com
5. For unknown primary or known primary not included within brainmetgpa.com, an estimated median survival no less than 6 months per PI discretion Note: If patient's estimated median survival is calculated using a histology that is different than the histology demonstrated in final pathology, the patient may remain eligible for all study endpoints per PI discretion
6. Surgical candidate per neurosurgeon discretion
7. Surgical resection able to be performed within 1 - 4 days after radiosurgery
8. Stereotactic radiosurgery candidate per radiation oncologist
9. ≥ 18 years old at the time of informed consent
10. Ability to provide written informed consent and HIPAA authorization. This will be assessed by the consenting physician using general questions to determine the patient's ability to understand the medical problem, proposed treatment, alternatives to proposed treatment, and understand the consequences of the medical choices.
11. Platelet count > 100 k/cumm, Hgb > 7.5 gm/dL, INR < 1.3, ANC > 1.5 k/cumm
12. Patients currently on cytotoxic chemotherapy or immunotherapy are eligible, not including anti-VEGF therapy
13. If a patient who meets all stated eligibility criteria is enrolled on study and then discovered to be ineligible, the tissue obtained will still be deemed eligible to remain in study for evaluation.

Exclusion Criteria

1. Patients who received anti-VEGF therapy within 6 weeks prior to enrollment, as there is increased risk of fatal brain hemorrhage with surgical resection
2. Major medical illnesses or psychiatric impairments, which in the investigator's opinion will prevent administration or completion of the protocol therapy and/or interfere with follow-up
3. Patients with more than 4 brain metastases on MRI Brain or CT Head
4. Lesion to be resected is more than 5 cm
5. Total volume of metastatic disease more than 30 cm3 excluding lesion to be resected
6. Patients with leptomeningeal metastases documented by MRI or CSF evaluation
7. Previous whole brain radiation therapy
8. Previous radiation therapy to lesion to be resected
9. Planned adjuvant focal therapy including additional radiation therapy to the brain
10. Not a surgical candidate per neurosurgeon's discretion
11. Not a radiosurgical candidate per radiation oncologist's discretion
12. Surgery unable to be performed between 1 - 4 days after radiosurgery
13. Women who are pregnant or nursing are not eligible as treatment involves unforeseeable risks to the fetus or child

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Rate of local control of any new, recurrent, or progressing tumors within the planning target volume | 6 months
  Measured by post-treatment MRI

SECONDARY OUTCOMES:
Rate of overall survival | 6 months, 1 year, and 2 years
  Time from start of treatment to death of any cause
Rate of in-brain progression free survival | 6 months, 1 year, and 2 years
  Time from start of treatment to any in-brain
Proportion of patients with distant in-brain failure (any new parenchymal lesion outside of the planning target volume) | 2 years
  Measured by post-treatment MRI
Proportion of patients with radiation necrosis (radiographic or biopsy-positive diagnosis of radiation necrosis) | 2 years
  Measured by post-treatment MRI
Proportion of patients with leptomeningeal spread (radiographic or CSF diagnosis of leptomeningeal disease) | 2 years
  Measured by post-treatment MRI

OTHER OUTCOMES:
Exploratory: Correlation of RNA biomarkers | 2 yrs
  Correlation of RNA biomarkers with local control

CONTACTS AND LOCATIONS:
Overall Officials: Namita Agrawal, MD, Principal Investigator — Indiana University School of Medicine
Locations (3):
- United States (3):
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huff WX, Agrawal N, Shapiro S, Miller J, Kulwin C, Shah M, Savage JJ, Payner T, Vortmeyer A, Watson G, Dey M. Efficacy of pre-operative stereotactic radiosurgery followed by surgical resection and correlative radiobiological analysis for patients with 1-4 brain metastases: study protocol for a phase II trial. Radiat Oncol. 2018 Dec 20;13(1):252. doi: 10.1186/s13014-018-1178-8. PMID 30572923